CLINICAL TRIAL: NCT06202222
Title: Interest of Intensive Postoperative Rehabilitation Following Minimally Invasive Lung Resection: A Randomized Controlled Study
Brief Title: Interest of Intensive Postoperative Rehabilitation Following Minimally Invasive Lung Resection
Acronym: IRPOL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020/0427/HP
Record Dates: First submitted 2023-12-29; First posted 2024-01-11 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard rehabilitation (No Intervention)
- standard rehabilitation and cycloergometer (Experimental)
  Interventions: Other: rehabilitation

INTERVENTIONS:
Other: rehabilitation — The patient undergoes a daily session on the cycloergometer (Am3i Ergometer). The patient is instructed to pedal at a heart rate ranging from 60% to 80% of their maximum heart rate (calculated as 220 minus their age) for a duration of 20 minutes. These sessions can be conducted with oxygen therapy for patients dependent on oxygen. The sessions are maintained until the patient is discharged from the department.
  Arms: standard rehabilitation and cycloergometer

SUMMARY:
For patients diagnosed with non-small cell lung cancer (NSCLC), lung resection surgery remains the gold standard for curative treatment. This scheduled operation is associated with significant morbidity, particularly in individuals with impaired cardio-respiratory function. Therefore, patient optimization is paramount. The process begins prior to surgery with preoperative rehabilitation, commonly referred to as "prehabilitation," serving as the foundation for various Enhanced Recovery After Surgery programs. The training methods employed in these programs bear similarity to rehabilitation programs designed for patients with chronic obstructive pulmonary disease (COPD).

Postoperatively, patients undergoing thoracic surgery partake in daily physiotherapy sessions, aiming to optimize the postoperative period, minimize the respiratory impact of surgery, and reduce the length of hospital stay. However, this treatment is not currently standardized and primarily involves early mobilization, including walking, and respiratory physiotherapy. Our focus is on the intensity and methods of this postoperative rehabilitation.

There is limited literature on effective early rehabilitation in the immediate postoperative period, and existing studies suggest no adverse events associated with postoperative training. Therefore, our objective is to assess whether combining endurance training with standard physiotherapy (walking and respiratory physiotherapy) enhances the functional capacity of individuals undergoing lung surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring surgery for diagnosed or undergoing diagnosis of lung cancer.
* Patients in need of major lung resection through a minimally invasive approach.
* Patients capable of performing the chair rise test.

Exclusion Criteria:

- Contraindications to cyclo-ergometry: Deep vein thrombosis in a lower limb. Patients with one or both lower limbs amputated. Rheumatological pathology, trauma, or previous surgery in the lower limb, pelvis, or spine, resulting in limited joint amplitude or strict immobilization.

Dermatological conditions with severe lesions preventing prolonged sitting on a bicycle.

* Glasgow score less than 15.
* Patients who have not undergone pulmonary resection by minimally invasive surgery.
* Patients hospitalized outside the thoracic surgery department before the first post-operative visit with the physiotherapist on Day 0.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2024-09-09 (Actual); Primary Completion 2027-05-09 (Estimated); Study Completion 2027-05-09 (Estimated)

PRIMARY OUTCOMES:
Number of chair lifts at the scheduled visit 30 days after surgery | 30 days after surgery
  number of chair lifts

SECONDARY OUTCOMES:
number of days between surgery and discharge patient | 30 days after surgery
chair rise test | 7 days after surgery
number of complication GRADE II of clavien dindo classification | 30 days after surgery

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Valenciennes, Hospital, Valenciennes, Hauts-de-France
  - CAEN, university Hospital, Caen, Normandy
  - Rouen, University Hospital, Rouen, Normandy

IPD SHARING:
Plan to Share IPD: No